CLINICAL TRIAL: NCT07344298
Title: Less is Better? Effectiveness of a Short Local Vibration Protocol on Neuromuscular Function
Acronym: VIB-EXPRESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25CH170; ANSM (Other: 2025-A01910-49)
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volonteers
Keywords: neuromuscular function; local vibration protocol; knee extensor

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, controlled trial comparing four groups of healthy volunteers following a protocol involving local vibration applied to the knee extensor muscles of the dominant leg. Two groups will follow a short-term intervention program consisting of 5 consecutive days of 30 or 60 minutes of vibration (5 sessions), while the other two will benefit from a program spread over 4 weeks at a rate of 3 sessions per week of 30 or 60 minutes of vibration (a total of 12 sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group "5 days and 30 min" (Experimental): Participants will follow a protocol involving local vibration applied to the quadriceps muscle for 5 consecutive days, at a rate of one 30-minute session per day.
  Interventions: Device: Local vibration protocol
- Group "5 days and 60 min" (Experimental): Participants will follow a protocol involving local vibration applied to the quadriceps muscle for 5 consecutive days, at a rate of one 60-minute session per day.
  Interventions: Device: Local vibration protocol
- Group "4-weeks and 30 min" (Experimental): Participants will follow a protocol involving local vibration applied to the quadriceps muscle over a period of 4 weeks, with 3 weekly sessions of 30 minutes each, for a total of 12 sessions.
  Interventions: Device: Local vibration protocol
- Group "4-weeks and 60 min" (Experimental): Participants will follow a protocol involving local vibration applied to the quadriceps muscle over a period of 4 weeks, with 3 weekly sessions of 60 minutes each, for a total of 12 sessions.
  Interventions: Device: Local vibration protocol

INTERVENTIONS:
Device: Local vibration protocol — The vibrations will be delivered using the Vibramoov Physio device, positioned directly on the quadriceps muscle. The participant will be seated comfortably and will remain at rest throughout the session. The vibration settings will be set to an amplitude of 1 mm and a frequency of 100 Hz.
  Other Names: Vibramoov Physio

SUMMARY:
Local vibration is a non-invasive neuromuscular stimulation modality used in training and rehabilitation for its effects on neuromuscular function, particularly its ability to induce nervous adaptations. Its passive application is particularly useful in cases of motor deficit or immobilization.

Several studies, including our own, have shown that vibration protocols over several weeks can induce significant gains in muscle strength, particularly in the knee extensors. However, the parameters of application remain heterogeneous, particularly with regard to the duration of the interventions.

With this in mind, a prospective controlled study is being conducted in healthy subjects, comparing four modalities of local vibration intervention targeting the knee extensors: an intensive vibration protocol over 5 consecutive days (1 session of 30 or 60 minutes per day) and a protocol spread over 4 weeks at a rate of 3 weekly sessions of 30 or 60 minutes). The objective is to evaluate and compare their immediate and delayed effects on force production and corticospinal properties. The results of this study will thus help optimize recommendations regarding the use of local vibration in muscle strengthening and neuromuscular reconditioning strategies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women,
* Aged between 18 and 45,
* With a body mass index between 20 and 25 kg/m²,
* Who have received detailed information about the study and have co-signed the consent form with the investigator,
* Who are affiliated with or entitled to social security coverage.

Exclusion Criteria:

* Subjects with chronic cardiovascular, neuromuscular, bone, metabolic, and/or inflammatory conditions,
* Personal history and/or risk factors for thrombosis,
* Subjects undergoing antidepressant treatment,
* Subjects who have taken corticosteroid treatment in the last 3 months,
* Use of neuroactive substances likely to alter corticospinal excitability (hypnotics, antiepileptics, psychotropic drugs, muscle relaxants) during the study period,
* History of bone or ligament trauma to the lower limbs within the last 12 months,
* Unable to perform the physical efforts required for the study,
* Engaging in intense and unusual physical activity, including competitive sports, in the month preceding and during the protocol,
* Presence of a skin lesion at the site where the vibrator is to be placed,
* Simultaneous participation in another interventional medical trial,
* Pregnant and breastfeeding women
* Subjects unable to understand the purpose and conditions of the study, unable to give their consent,
* Subjects deprived of their liberty or subject to legal protection such as guardianship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on the gain in knee extension strength in healthy volunteers. | Five times: before the procedure (baseline); at the end of the procedure (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70), and 3 months (day 105 or day 126) after the procedure.
  The primary endpoint will be the relative change in maximum isometric strength of the knee extensors (expressed as a percentage increased), assessed using an isokinetic dynamometer.

SECONDARY OUTCOMES:
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on functional motor abilities and, more specifically, maximum voluntary strength | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  Strength (Nm) will be assessed on an isokinetic dynamometer. Two concentric contraction speeds will be tested: 60°/s and 180°/s (also assessed for the contralateral leg).
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on functional motor skills and, more specifically, jumping performance. | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  Jumping performance (height, in cm) will be assessed using validated vertical jump tests: Squat Jump and Counter Movement Jump.
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on functional motor skills and, more specifically, the rate of force development (RFD) | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  The RFD (expressed in N/s), an indicator of explosive strength, will be assessed for the knee extensor muscles from the initial phases of isometric contraction on an isokinetic dynamometer.
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on corticospinal properties and, more specifically, on the level of voluntary activation | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  The level of voluntary activation (in %) will be determined by the increase in force obtained following electrical nerve stimulation during a maximum voluntary isometric contraction. An electrical stimulator will deliver rectangular electrical pulses (400 V max, pulse duration: 1 ms) to the femoral nerve through the skin.
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on corticospinal properties and, more specifically, corticospinal excitability. | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  Cortico-spinal excitability will be assessed using electromyographic responses (motor evoked potentials, in mV) elicited by transcranial magnetic stimulation.
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on corticospinal properties and, more specifically, spinal excitability | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  Spinal excitability (in mV) will be assessed by recording electromyographic responses evoked by electrical stimulation at the femoral nerve and spinal cord (thoracic motor evoked potentials).
Compare the effect of the duration of a local vibration program (5 days vs 4 weeks), as well as the effect of the duration of the sessions (30 min vs 60 min) on corticospinal properties and, more specifically, cortical activation of sensorimotor areas. | Five times: before the intervention (baseline); at the end of the intervention (day 21 or day 42 depending on the group); then 1 week (day 28 or day 49), 1 month (day 49 or day 70) and 3 months (day 105 or day 126) after the intervention.
  Cortical activation of sensorimotor areas will be assessed by recording the electroencephalographic signal during submaximal isometric contractions. A flexible 64-electrode cap will be placed on the subject's head and a gel will be applied to improve signal reception. The signal will be recorded at rest during a 3-minute period of muscle inactivity, then during a 30-minute vibration session.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD, PhD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No